CLINICAL TRIAL: NCT05889533
Title: Increasing PrEP Options for Women in Eswatini: A Prospective Mixed Methods Study on the Introduction of the PrEP Vaginal Ring
Brief Title: Eswatini Ring Study: Increasing PrEP Options for Women
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to the stop work order issued by USAID on January 27, 2025
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FHI 360
Record Dates: First submitted 2023-05-26; First posted 2023-06-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: HIV Prevention
Keywords: HIV prevention; PrEP; AGYW; PrEP Ring; Eswatini

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will deliver PrEP choice between oral PrEP and the PrEP ring for women in PEPFAR/USAID public health service delivery sites, building on the existing PrEP service delivery models at each site and in accordance with national guidelines for PrEP service delivery in Eswatini. The overall goal of the study is to characterize and assess the feasibility, acceptability, uptake, patterns of use, and clinical outcomes of an enhanced service delivery package providing fully informed choice of oral PrEP and the PrEP ring among women, especially adolescent girls and young women, in Eswatini.

DETAILED DESCRIPTION:
The study will deliver PrEP choice between oral PrEP and the PrEP ring for women in PEPFAR/USAID public health service delivery sites, building on the existing PrEP service delivery models at each site and in accordance with national guidelines for PrEP service delivery in Eswatini. The overall goal of the study is to characterize and assess the feasibility, acceptability, uptake, patterns of use, and clinical outcomes of an enhanced service delivery package providing fully informed choice of oral PrEP and the PrEP ring among women, especially adolescent girls and young women, in Eswatini.

The two main study components include the following:

1. Prospective, observational cohort of eligible individuals interested in initiating PrEP or continuing PrEP with screening for entry at time of HIV testing and followed throughout the study period (up to 18 months). Data collection will involve quantitative methods and for a subset of participants, data will also be collected using qualitative means, namely in-depth interviews, and focus group discussions.
2. Mixed methods process evaluation that will document implementation of the enhanced service delivery package, assess ongoing perceptions of service delivery (i.e., acceptability and feasibility, barriers and facilitators) among providers and end users, and document other important implementation considerations including the integration of PrEP and family planning.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative, 18 or older, not known to be pregnant or breastfeeding, and female at birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Those meeting eligibility criteria seeking PrEP services at study sites.
Sampling Method: Non-Probability Sample
Enrollment: 904 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Characterize implementation of the service delivery package for informed PrEP choice for women | 18 months
  Health system feasibility and delivery acceptance among users/providers

SECONDARY OUTCOMES:
Describe patterns of PrEP use in the context of informed PrEP choice | 18 months
  Overall and method-specific PrEP uptake; continuation/switching/discontinuation of PrEP products; product acceptability among users.

OTHER OUTCOMES:
Describe clinically relevant indicators among PrEP users, including rates of seroconversion and drug resistance among PEP users who acquire HIV following PrEP initiation. | 18 months
  Proportion and rates of HIV infection among participants; proportion and rates of HIV drug resistance (DR) mutations among PrEP users who acquire HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Hettema, MPH, Principal Investigator — FHI 360; Sindy Matse, MPH, Principal Investigator — Ministry of Health
Locations (8):
- Eswatini (8):
  - Dvokolwako Health Centre, Dvokolwako
  - Manzini KP Community Centre, Manzini
  - Matsapha Mobile Clinic, Matsapha
  - Mbabane Key Population (KP) Community Centre, Mbabane
  - Mbabane Public Health Unit, Mbabane
  - Motshane Clinic, Mbabane
  - Siphofaneni Inkhundla (DREAMS Outreach), Siphofaneni
  - New Haven Clinic, Velebantfu

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the USAID Automated Directives System 579, after acceptance of any knowledge product presenting study findings and after being cleaned of any information that could be used to personally identify participants, the quantitative survey dataset along with relevant documentation will be registered with USAID's Development Data Library (DDL) and made available publicly in an open data repository, to the extent permissible by Eswatini's data privacy and data sharing regulations.
Supporting Information: Study Protocol, ICF
Time Frame: After study completion and manuscript submission.